CLINICAL TRIAL: NCT02882802
Title: Mindfulness Treatment for Anger in Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLNA-006-15F
Record Dates: First submitted 2016-07-22; First posted 2016-08-30 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Anger; Aggression
Keywords: anger; aggression
MeSH Terms: conditions — Aggression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): Mindfulness Based Stress Reduction (MBSR) is a group-based intervention in which participants are taught different mindfulness meditation practices, including body scan (focusing attention to different areas of the body in sequence), sitting meditation (focusing attention to one's breathing), and Hatha yoga postures (focusing attention to different body sensations during gentle stretching). Participants also are taught how to practice mindfulness while engaging in ordinary activities including walking, standing, and eating. MBSR consists of 8, two-hour weekly sessions and will be delivered in group format. MBSR groups will be delivered virtually.
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Trauma Recovery Education Class (Active Comparator): Trauma Recovery Education Class (TREC): TREC is a group based treatment that focuses on providing information on PTSD and traumatic reactions. TREC provides psycho-education to Veterans on PTSD, including common reactions to trauma and the role of avoidance, common problems associated with PTSD, as well as common barriers to care (e.g., stigma, maladaptive beliefs, fear). Additional content focuses on problem identification and goal setting, discussion of current problems and life issues, and treatment planning. TREC consists of 8, one-hour weekly sessions. TREC groups will be delivered virtually.
  Interventions: Behavioral: Trauma Recovery Education Class

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction — Mindfulness Based Stress Reduction (MBSR) is a group-based intervention in which participants are taught different mindfulness meditation practices, including body scan (focusing attention to different areas of the body in sequence), sitting meditation (focusing attention to one's breathing), and Hatha yoga postures (focusing attention to different body sensations during gentle stretching). Participants also are taught how to practice mindfulness while engaging in ordinary activities including walking, standing, and eating. MBSR consists of 8, two-hour weekly sessions and will be delivered in group format. MBSR groups will be delivered virtually.
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction
Behavioral: Trauma Recovery Education Class — Trauma Recovery Education Class (TREC): TREC is a group based treatment that focuses on providing information on PTSD and traumatic reactions. TREC provides psycho-education to Veterans on PTSD, including common reactions to trauma and the role of avoidance, common problems associated with PTSD, as well as common barriers to care (e.g., stigma, maladaptive beliefs, fear). Additional content focuses on problem identification and goal setting, discussion of current problems and life issues, and treatment planning. TREC consists of 8, one-hour weekly sessions. TREC groups will be delivered virtually.
  Other Names: TREC
  Arms: Trauma Recovery Education Class

SUMMARY:
Research has consistently shown that Veterans with PTSD are more likely to experience higher levels of anger and commit aggressive acts compared to Veterans without PTSD. Given the significant negative impact that anger and aggression can have on the lives of Veterans, their families, and society at large, there is a great need to examine novel interventions that could decrease anger and aggression risk with this population. Mindfulness may be one such technique, given its effectiveness in assisting individuals in regulating difficult emotions and in decreasing physiological reactivity, which have both been implicated in PTSD and aggression perpetration. Findings showing that a mindfulness intervention is effective in reducing anger and aggressive behavior would be relevant for Veterans with PTSD experiencing such difficulties and would help prevent the detrimental consequences that can come from anger and aggression among these individuals.

DETAILED DESCRIPTION:
Military Veterans suffering from posttraumatic stress disorder (PTSD) have been shown to exhibit increases in aggressive urges, difficulties managing anger, and difficulties controlling violent behavior. Dysregulated anger and aggression can create fear and distress in spouses, family members, and friends resulting in strained and deteriorated relationships, and can have a detrimental impact on Veterans' social, occupational and other important areas of functioning. In addition, more severe forms of aggression and violent behavior (i.e., homicide) in the community have been observed among Veterans with PTSD, as recently reported in several news media outlets. The seriousness of this problem is underscored by the high rates of alcohol use observed among Veterans with PTSD which further increases anger and the risk of aggressive behavior.

Current therapeutic interventions may not be effective in reducing anger and aggressive behavior among Veterans with PTSD due to the lack of techniques that directly target symptoms most strongly associated with aggression, particularly hyperarousal and physiological reactivity. Furthermore, existing interventions may not be effective in assisting individuals achieve awareness and insight into their anger states, necessary for the effective management of anger and aggression. Mindfulness is rooted in Eastern meditation practices and has been successfully used to decrease stress, pain, anxiety, and depression. In civilian samples, mindfulness interventions have been found to be effective in reducing anger and aggression. To date, mindfulness for anger and aggression has not been examined in Veterans with PTSD.

The primary objective of the proposed investigation is to conduct a pilot randomized control trial to examine the initial efficacy of an established mindfulness intervention, Mindfulness Based Stress Reduction (MBSR) in decreasing anger and aggression in Veterans with PTSD. The proposed investigation also seeks to examine potential mechanisms of action that account for its effects. Sixty Veterans with PTSD experiencing problems with anger and aggression will be recruited. These individuals will complete a baseline assessment to assess self-reported levels of anger and aggression. They will then be randomly assigned to participate in an online (i.e., virtual) PTSD psychoeducational course or MBSR. After completing treatment, all participants will complete a post-treatment assessment to assess changes in anger and aggression.

At a later date and time, participants will also be asked to attend an in-person laboratory session where they will engage in a trauma-imagery procedure followed by a task designed to assess provoked aggression. In addition to examining whether participation in MBSR decreases self-reported levels of anger and aggression, this study will examine whether MBSR decreases aggression in participants after being exposed to trauma reminders in vivo. Potential mechanisms of action of MBSR and its effects on additional outcomes also will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet current DSM-V diagnostic criteria for PTSD (participants with sub-threshold levels of PTSD will also be allowed to participate).
* Participants must also indicate current difficulties with anger and aggression.

Exclusion Criteria:

* Participants with a current diagnosis of psychotic disorder or current substance use disorder with severe symptoms.
* Participants diagnosed with bipolar II disorder without psychotic features and/or individuals diagnosed with bipolar disorder who are well-controlled on medication will be allowed to participate. Individuals with bipolar disorder who do not fall into either of these categories will be excluded.
* Participants also must not have a seizure disorder.
* Participants are allowed to be taking psychotropic medications, however they must be on a stable dose for at least 2 months.
* Participants who do not have a working and active e-mail account and access to a smartphone or computer will be excluded.
* Finally, participants must not currently be receiving concurrent individual therapy or group therapy focused on anger and aggression, must not be currently receiving any evidence-based treatment for PTSD, and must not currently be participating in the modified TREC group offered at the WHVA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
anger | Baseline, after 3 weeks of treatment, within 4 weeks following the completion of either of the two treatments, after 6 weeks of treatment, 3-month follow up
  changes in a self report measure of anger using the State-Trait Anger Expression Inventory-2
aggression | Baseline, after 3 weeks of treatment, within 4 weeks following the completion of either of the two treatments, after 6 weeks of treatment, 3-month follow up
  changes in a self report measure of aggression using the Buss-Perry Aggression Questionnaire
provoked aggression | within 4 weeks following the completion of either of the two treatments
  An experimental lab-based paradigm designed to assess provoked aggression, the Taylor Reaction Time Task

SECONDARY OUTCOMES:
heart rate | within 4 weeks following the completion of either of the two treatments
  physiological assessment implemented while participants are exposed to trauma narratives
skin-conductance levels | within 4 weeks following the completion of either of the two treatments
  physiological assessment implemented while participants are exposed to trauma narratives

CONTACTS AND LOCATIONS:
Overall Officials: Lorig Kachadourian, PhD MA, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No